CLINICAL TRIAL: NCT03706898
Title: Open Label Study to Evaluate the Safety and Pharmacokinetics of Elpida® in Healthy Subjects and Patients With Hepatic Impairment, as Well as to Assess the Impact of Food Intake and Drug-Drug Interactions in Case of Co-administration With Other Antiviral Drugs in Healthy Subjects
Brief Title: Study to Evaluate the Safety and PK of Elpida® in Healthy Subjects and Patients With Hepatic Impairment and to Assess the Impact of Food Intake and Drug-Drug Interactions With Other Antiviral Drugs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viriom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HIV-VM1500-07
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2020-05

CONDITIONS: HIV-1-infection; Hepatic Impairment
MeSH Terms: interventions — elsulfavirine; dolutegravir; Sofosbuvir; daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Elpida® fasting (Experimental): Elpida® 20 mg single dose fasting
  Interventions: Drug: Elpida®
- Elpida® after meal (Experimental): Elpida® 20 mg single dose after meals
  Interventions: Drug: Elpida®
- Elpida® (in subjects with mild hepatic impairment) (Experimental): Elpida® 20 mg single dose fasting - subjects with mild hepatic impairment (Child - Pugh Class А)
  Interventions: Drug: Elpida®
- Elpida® (in subjects with moderate hepatic impairment) (Experimental): Elpida® 20 mg single dose fasting - subjects with moderate hepatic impairment (Child - Pugh Class B)
  Interventions: Drug: Elpida®
- Elpida® & sofosbuvir & daclatasvir (Experimental): Drug-drug interactions of sofosbuvir 400 mg + daclatasvir 60 mg and Elpida® 20 mg, single dose fasting
  Interventions: Drug: Elpida®; Drug: Sofosbuvir; Drug: Daclatasvir
- Elpida® & dolutegravir (Experimental): Drug-drug interactions of dolutegravir 50 mg and Elpida® 20 mg, single dose fasting
  Interventions: Drug: Elpida®; Drug: Dolutegravir

INTERVENTIONS:
Drug: Elpida® — Elpida® capsules, 20mg
  Other Names: Elsulfavirine; VM1500; VM-1500
Drug: Dolutegravir — Dolutegravir, film-coated tablets, 50mg
  Other Names: TIVICAY®
  Arms: Elpida® & dolutegravir
Drug: Sofosbuvir — Sofosbuvir, film-coated tablets, 400mg
  Other Names: Sovaldi
  Arms: Elpida® & sofosbuvir & daclatasvir
Drug: Daclatasvir — Daclatasvir, film-coated tablets, 60mg
  Other Names: Daklinza®
  Arms: Elpida® & sofosbuvir & daclatasvir

SUMMARY:
This is open label, phase 1 clinical study to evaluate the safety, tolerability and pharmacokinetics of Elpida® in healthy subjects and patients with hepatic impairment (Child - Pugh Class А and B), as well as to assess the impact of food intake and drug-drug interactions in case of Co-administration with other antiviral drugs in healthy subjects.

DETAILED DESCRIPTION:
In medical practice HIV infection is often found associated with viral hepatitis, especially chronic hepatitis C virus (HCV). This, as well as a possible change in PK parameters in case of co-administration of Elpida® and HIV integrase inhibitors, necessitates the study of PK and safety of co-administration of Elpida® with a combination of Sofosbuvir + Daclatasvir and Dolutegravir in healthy subjects. Thus, the study to evaluates safety and pharmacokinetics of Elpida® in healthy subjects and patients with hepatic impairment, as well as assesses the impact of food intake and drug-drug interactions in case of co-administration with other antiviral drugs in healthy subjects.

ELIGIBILITY:
Inclusion Criteria for healthy volunteers:

1. Non-smoking male or female subjects between the ages of 18 and 45 years (inclusive);
2. Verified "healthy" diagnosis according to standard clinical, laboratory and instrumental examination methods;
3. Body Mass Index ranges between 18.5 kg/m2 and 30.0 kg/m2 and a body weight not less than 50 kg;
4. Negative alcohol and drug tests;
5. Consent to use two adequate and reliable methods of contraception throughout the study and up to 3 months after its completion: a condom with spermicide (foam, gel, cream, suppositories), or a diaphragm with spermicide, or a condom and diaphragm, or a condom and an intrauterine device;
6. Signed Patient Information Sheet and form of Informed Consent to participate in the study.

Inclusion Criteria for patients with hepatic impairment:

1. Non-smoking male or female subjects between the ages of 18 and 45 years (inclusive);
2. Mild and moderate hepatic impairment (Child - Pugh Class A or B), including viral nature (Hepatitis C virus, etc.). At the same time, there were no changes in the diagnosis of the patient according to Child - Pugh Class not less than 1 month prior to screening;
3. Increase in the concentration of aspartate aminotransferase (AST )and (or) alanine aminotransferase (ALT) in blood plasma by 1.25 times or more from the upper limit of the norm (ULN), but not more than 5 times ULN at the time of screening;
4. Body Mass Index ranges between 18.0 kg/m2 and 36.0 kg/m2 and a body weight not less than 50 kg, but not more than 120 kg;
5. Negative alcohol and drug tests;
6. Consent to use two adequate and reliable methods of contraception throughout the study and up to 3 months after its completion: a condom with spermicide (foam, gel, cream, suppositories), or a diaphragm with spermicide, or a condom and diaphragm, or a condom and an intrauterine device;
7. Signed Patient Information Sheet and form of Informed Consent to participate in the study.

Exclusion Criteria:

1. Chronic diseases of cardiovascular, bronchopulmonary, neuroendocrine, musculoskeletal system, as well as diseases of the gastrointestinal tract, liver, kidneys, blood;
2. Variables of standard laboratory and instrumental parameters are beyond the normal limits (taking into account the acceptable limits of laboratory parameters);
3. Surgical interventions on the gastrointestinal tract in medical history (except appendectomy);
4. Systolic pressure below 90 mmHg or above 130 mmHg, diastolic pressure below 60 mmHg or above 85 mmHg, heart rate less than 60 BPM or more than 90 BPM at screening;
5. Regular intake of drugs less than 2 weeks prior to screening (including herbal preparations and dietary supplements); intake of drugs that have a pronounced effect on hemodynamics, hepatic function, etc. (for example, barbiturates, omeprazole, cimetidine, etc.) less than 30 days prior to screening;
6. Presence of antibodies to HIV and hepatitis C virus, presence of hepatitis В surface antigen, a positive syphilis test;
7. An unstable sleep structure (e.g., night work, sleep disorders, insomnia, recent return from another time zone, etc.), extreme physical activity (e.g. weight lifting), a special diet (e.g. vegetarian, vegan);
8. Signs of alcohol (intake of more than 10 units of alcohol per week ) or drug addiction; alcohol or drugs consumption within 4 days prior to screening; cigarettes smoking 3 months prior to screening; positive drug and/or alcohol test;
9. Drug allergies in medical history (including drug intolerance, including hypersensitivity to active / excipient substances of study drugs - elsulfavirine, sofosbuvir, daclatasvir, dolutegravir as well as any other substance of study drugs ) as well as food allergy;
10. Lactase deficiency, lactose intolerance, glucose-galactose malabsorption;
11. Blood/plasma donation (450 ml of blood or plasma and more) less than 2 months prior to screening;
12. Participation in other clinical studies or taking other study drugs 1 months prior to screening;
13. Acute infectious diseases less than 4 weeks prior to screening;
14. Inhibitors or inducers of CYP3A4/5, drugs that cause QTс prolongation () within 30 days prior to Study Drug administration;
15. For women - positive result of pregnancy test or breastfeeding;
16. Inability to read or write; unwillingness to understand and adhere to the study protocol procedures; non-compliance with the drugs intake regimen or execution of procedures, which as the Investigator believes may affect the study results or subject's safety and prevent the subject from further participation in the study; any other associated medical or serious psychological conditions making the subject not eligible to participate in the clinical study, restricting legality of obtaining the Informed Consent or affecting the subject's ability to participate in the study.

Exclusion criteria for patients with hepatic impairment:

1. Severe hepatic impairment (Child - Pugh Class C); other hepatic disorders or conditions that do not allow according to the Investigator to include the patient in the study without increased threat to his safety - including (but not limited to) signs of severe ascites requiring regular abdominal laparocentesis, the level of total bilirubin in blood plasma > 100 µmol/l, etc.;
2. Chronic diseases of cardiovascular, bronchopulmonary, neuroendocrine, musculoskeletal system, as well as diseases of the gastrointestinal tract, kidneys, blood, requiring medical treatment and preventing, according to the Investigator the subject's participation in the study;
3. Surgical interventions on the gastrointestinal tract in medical history including liver transplantation (except appendectomy);
4. Regular intake of drugs less than 2 weeks prior to study drug administration (including herbal preparations and dietary supplements); intake of drugs that have a pronounced effect on hemodynamics, hepatic function, etc. (for example, barbiturates, omeprazole, cimetidine, etc.) less than 30 days prior to study drug administration;
5. Antibodies to HIV, a positive syphilis test;
6. An unstable sleep structure (e.g., night work, sleep disorders, insomnia, recent return from another time zone, etc.), extreme physical activity (e.g. weight lifting), a special diet (e.g. vegetarian, vegan);
7. Signs of alcohol (taking more than 10 units of alcohol per week) or drug addiction; alcohol or drugs consumption within 4 days prior to screening; cigarettes smoking 3 months prior to screening; positive drug and/or alcohol test;
8. Drug allergies in medical history (including drug intolerance, including hypersensitivity to active / excipient substances of Elpida®) as well as food allergy;
9. Lactase deficiency, lactose intolerance, glucose-galactose malabsorption;
10. Participation in other clinical studies or taking other study drugs 1 months prior to screening;
11. Acute infectious diseases less than 4 weeks prior to screening;
12. Any prescribed pharmacotherapy aimed at restoring hepatic function, eradication of hepatitis viruses, or otherwise focused on the compensation of hepatic impairment;
13. Administration of inhibitors or inducers of CYP3A4/5, drugs that cause QTс prolongation within 30 days prior to StD administration; ongoing therapy with immunosuppressive agents;
14. For women - positive result of pregnancy test or breastfeeding;
15. Inability to read or write; unwillingness to understand and adhere to the study protocol procedures; non-compliance with the drugs intake regimen or execution of procedures, which as the Investigator believes may affect the study results or subject's safety and prevent the subject from further participation in the study; any other associated medical or serious psychological conditions making the subject not eligible to participate in the clinical study, restricting legality of obtaining the Informed Consent or affecting the subject's ability to participate in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of elsulfavirine | 42 days
Plasma concentration of VM-1500A | 42 days
Plasma concentration of daclatasvir | 42 days
Plasma concentration of sofosbuvir | 42 days
Plasma concentration of dolutegravir | 42 days

SECONDARY OUTCOMES:
AEs and SAEs frequency | 42 days
  Adverse events (AE) and serious adverse events (SAE) frequency of varying severity according to subjective complaints, physical examination, instrumental and laboratory studies

CONTACTS AND LOCATIONS:
Overall Officials: Alla Andreeva, PhD, Principal Investigator — Regional State Budgetary Healthcare Institution "Smolensk Regional Clinical Hospital"
Locations (1):
- Regional State Budgetary Healthcare Institution "Smolensk Regional Clinical Hospital", Smolensk, Russia

IPD SHARING:
Plan to Share IPD: No